CLINICAL TRIAL: NCT05861505
Title: COLLISION RELAPSE Trial - Recurrent Colorectal Liver Metastases: Repeat Local Treatment +/- Neoadjuvant Systemic Therapy - a Phase III Prospective Randomized Controlled Trial
Brief Title: COLLISION RELAPSE Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.R. Meijerink, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL78220.029.21
Record Dates: First submitted 2023-04-26; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Liver Metastases; Liver Metastasis Colon Cancer; Chemotherapy Effect; Surgery; Recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront repeat local treatment (Active Comparator)
  Interventions: Other: Repeat local treatment
- Neoadjuvant systemic therapy followed by repeat local treatment (Experimental)
  Interventions: Drug: Neoadjuvant systemic therapy (CAPOX+/-B FOLFOX+/-B FOLFIRI+/-B); Other: Repeat local treatment

INTERVENTIONS:
Drug: Neoadjuvant systemic therapy (CAPOX+/-B FOLFOX+/-B FOLFIRI+/-B) — Standard first line systemic treatment:
  CAPOX+/-B FOLFOX+/-B FOLFIRI+/-B
  CAPOX 4x (12 weeks) FOLFOX/FOLFIRI 6x (12 weeks)
  Maximum 4 cycles of CAPOX or 6 cycles of FOLFOX/FOLFIRI +/- bevacizumab regardless of the location of primary tumor or RAS/BRAF mutation
  Arms: Neoadjuvant systemic therapy followed by repeat local treatment
Other: Repeat local treatment — Choice of repeat local treatment is to the discretion of the local investigator, and may be selected on a per patient basis.
  The safety, feasibility and preferred type of surgical resection(s) is at the discretion of the liver surgeon (whether or not combined with thermal ablation).
  The safety, feasibility and preferred type of thermal ablation(s) is at the discretion of the interventional radiologist (whether or not combined with surgical resection).

SUMMARY:
The primary objective is to demonstrate superiority of neoadjuvant systemic therapy followed by repeat local treatment as compared to upfront repeat local treatment in patients with at least one locally treatable recurrent CRLM in the absence of extrahepatic disease.

DETAILED DESCRIPTION:
Study design: The COLLISION RELAPSE trial is a prospective multicenter phase III randomized controlled trial. The primary conducting center will be the Amsterdam UMC (Amsterdam, the Netherlands). We hypothesize that neoadjuvant systemic therapy followed by repeat local treatment is superior to upfront repeat local treatment for the selected patient groups in terms of the primary objective (OS). The Cox proportional hazards model (1-sided; superiority) and the PASKWIL criteria for adjuvant treatment for the benefit of OS from the Dutch Society of Medical Oncology are used for the sample size calculations. A total number of 360 patients will be randomized (NR) into one of two arms: arm A (control group) upfront repeat local treatment (n=180) and arm B (intervention group) 12 weeks of neoadjuvant systemic therapy followed by repeat local treatment (n=180).

Study population: Patients with a maximum of 5 recurrent new locally treatable CRLM within 12 months after initial curative intent local treatment of CRLM, no extrahepatic disease, and a good performance status (ECOG 0-2) are considered eligible. Both chemo-naïve patients and patients who did not progress on either oxaliplatin or irinotecan chemotherapy prior to the initial local treatment are eligible for inclusion.

Eligible patients will be stratified before randomization into two groups depending on the interval between initial local treatment and first detection of recurrent CRLM: recurrence within 6 months and recurrence between 6 and 12 months, RAS/BRAF mutation vs RAS/BRAF wildtype, prognostic risk score (low vs high risk, clinical risk score Fong et al. (83)) and previous chemotherapy versus no previous chemotherapy.

Intervention: Eligible patients will be randomized into one of two arms: arm A (control group) upfront repeat local treatment and arm B (intervention group) 12 weeks of neoadjuvant systemic therapy followed by repeat local treatment. Patients in arm B will receive maximum 4 cycles of CAPOX or 6 cycles of FOLFOX/FOLFIRI +/- bevacizumab regardless of the location of primary tumor or RAS/BRAF mutation. Choice of repeat local treatment is to the discretion of the local investigator, and may be selected on a per patient basis.

ELIGIBILITY:
Inclusion criteria

* Age >18 years
* Good performance status (ECOG 0-2 // ASA 1-3)
* Histological documentation of primary colorectal tumor
* Local treatment performed for initial CRLM
* New recurrence ≤12 months
* ≥1 locally treatable CRLM (resectable* and/or ablatable)
* Total number of new CRLM ≤5
* Chemo-naïve or history of response to CAPOX/FOLFOX/FOLRIRI
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function
* Written informed consent Exclusion criteria
* Extrahepatic disease
* MSI/dMMR
* Radical local treatment unfeasible or unsafe (e.g. insufficient future liver volume)
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites)
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0)
* Pregnant or breast-feeding subjects
* Immuno- or chemotherapy ≤ 6 weeks prior to the randomization
* Severe allergy to contrast media not controlled with premedication
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results

ECOG = Eastern Cooperative Oncology Group, ASA = American Society of Anesthesiologists, MSI = Microsatellite instability, dMMR = deficient mismatch repair

* Resection for resectable lesions considered possible obtaining negative resection margins (R0) and preserving adequate liver reserve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) per patient | 5 years
  Primary objective is to compare overall survival (OS) in both study arms, counting from the date of randomization to the date of death of the patient or to the last day of follow-up (censored).

SECONDARY OUTCOMES:
Distant progression-free survival (DPFS) per patient | 5 years
  Distant progression free survival (DPFS; per patient analysis): Overall DPFS is defined as the time from randomization to the time of disease progression (according to the RECIST 1.1 guideline) or cancer related death (events), death related to other causes is considered a competing risk
Local tumor progression-free survival (LTPFS) per patient and per tumor treated | 5 years
  Local tumor progression free survival (LTPFS; per tumor and per patient analysis): Overall LTPFS is defined as the time from randomization to the time of local disease progression, new metastases (events), censoring the date of death from any cause (competing risk), completion ablations performed within 6 weeks for residual tumor are not considered events for the local tumor progression analysis
Systemic therapy related toxicity per patient following neoadjuvant systemic therapy | 5 years
  Systemic therapy related toxicity is graded from 1 to 5 according to the CTCAE version 5.0
Procedural morbidity and mortality per patient following repeat local treatment | 5 years
  Procedural morbidity and mortality are graded from I to V according to the standard classification of surgical complications
Length of hospital stay per patient following repeat local treatment | 5 years
  In days
Assessment of pain per patient | 5 years
  - Pain assessment using visual analogue scale questionnaires (VAS; per procedure analysis: Assessed prior to, directly after and every three months after local treatment;
Quality of life (QoL) per patient | 5 years
  - To determine quality of life in both treatment arms. Quality of life assessment using EORCT QLQ-C30, EQ-5D, and PRODISQ questionnaires (per procedure analysis): Assessed prior to, and every three months after local treatment, assessed prior to, during and after neoadjuvant systemic therapy
Quality-adjusted life years (QALY) per patient | 5 years
  - Quality-adjusted life years (QALY) per treatment arm (per patient analysis).
Cost-effectiveness ratio (ICER) | 5 years
  - Direct and indirect total costs of care per treatment arm, and incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dijkstra M, Kuiper BI, Schulz HH, van der Lei S, Puijk RS, Vos DJW, Timmer FEF, Scheffer HJ, Buffart TE, van den Tol MP, Lissenberg-Witte BI, Swijnenburg RJ, Versteeg KS, Meijerink MR; COLLISION Trial Group. Recurrent Colorectal Liver Metastases: Upfront Local Treatment versus Neoadjuvant Systemic Therapy Followed by Local Treatment (COLLISION RELAPSE): Study Protocol of a Phase III Prospective Randomized Controlled Trial. Cardiovasc Intervent Radiol. 2024 Feb;47(2):253-262. doi: 10.1007/s00270-023-03602-y. Epub 2023 Nov 9. PMID 37943351